CLINICAL TRIAL: NCT00131547
Title: A Randomized Controlled Pilot Study of a Simple Weight Loss Program for Obese Patients With Mild to Moderate Obstructive Sleep Apnea
Brief Title: Randomized Study of a Simple Weight Loss Program for Obese Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Dr. Kathleen Ferguson, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-04-264; 10596
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obesity; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual Clinical Care
- 2 (Experimental): Behavioral (e.g., Counseling)
  Interventions: Behavioral: Dietary Counseling

INTERVENTIONS:
Behavioral: Dietary Counseling — Dietary Counseling, use of a food diary and pedometer
  Arms: 2

SUMMARY:
The purpose of the study is to determine if weight loss interventions aimed at lifestyle modification (dietary education, food diary pedometer) result in weight loss in patients with mild-moderate obstructive sleep apnea (OSA) when compared to usual patient care. The secondary purpose of the study is to determine if the amount of weight loss achieved in a 6 month period results in improvements in snoring and other symptoms and in the frequency of apnea on overnight monitoring.

DETAILED DESCRIPTION:
The purpose of the study is to determine if weight loss interventions aimed at lifestyle modification (dietary education, food diary pedometer) result in weight loss in patients with mild-moderate obstructive sleep apnea (OSA) when compared to usual patient care. The secondary purpose of the study is to determine if the amount of weight loss achieved in a 6 month period results in improvements in snoring and other symptoms and in the frequency of apnea on overnight monitoring.

Primary Objective

* To determine if weight loss interventions aimed at lifestyle modification (dietary education, food diary pedometer) result in weight loss in patients with mild-moderate OSA when compared to usual care.
* To determine if the amount of weight loss achieved in a 6 month period result in improvements in objective measures of sleep disordered breathing (AHI).

Secondary Objective

* To determine if the weight loss achieved in 6 months result in improvements in OSA symptoms (e.g., snoring, sleepiness) and quality of life.
* To determine if metabolic parameters (e.g., lipids, glucose) improve.
* To determine if there is improvement in sleep structure and oxygenation during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a sleep study at the London Health Sciences Centre or St. Thomas Elgin General Hospital Sleep Laboratory and who are newly diagnosed with obstructive sleep apnea
* Patients with an age over 18 years
* Patients who have an apnea-hypopnea index (AHI) of 5-40 per hour (mild-to-moderate OSA)
* Patients who have an elevated body mass index (BMI) of 28 to 39 kg/m2
* Patients who have an Epworth Sleepiness Scale score ≤11

Exclusion Criteria:

Patients will not be recruited:

* if they are on weight loss medications
* if they have seen a registered dietician in the preceding 6 months for dietary counseling
* if they have attended a weight loss program in the last 6 months
* if they have a history of a car accident related to sleepiness or report sleepiness when driving
* if they work in a safety critical occupation and require treatment for work reasons
* if they have serious or unstable cardiac co-morbidity
* if they are unable or unwilling to provide informed consent
* if they are pregnant
* if they are unwilling to return for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Post treatment weight (kg) | 6 months

SECONDARY OUTCOMES:
Change in snoring (Visual analogue scale) | 6 months
Quality of life (FOSQ) | 6 months
Excessive daytime sleepiness (ESS) | 6 months
Waist-hip ratio (WHR) | 6 months
Blood pressure | 6 months
Lipid and glucose levels | 6 months
Sleep fragmentation | 6 months
Oxygen saturation | 6 months
Post treatment AHI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ferguson, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada